CLINICAL TRIAL: NCT06187974
Title: Assessment of the Relationship Between the Deficit of Proprioception, Reaction Time and the Parameters of Gait and Balance in Stroke Patients
Brief Title: Relationship of Proprioception, Reaction Time and the Gait and Balance Parameters After Stroke
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Rzeszow (Other)
Responsible Party: Principal Investigator, Maciej Kochman, Principal Investigator, University of Rzeszow
Other Study IDs: Mkochman
Record Dates: First submitted 2023-07-03; First posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-12

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Study group: stroke patients
  Interventions: Other: observation
- Control group: healthy volunteers
  Interventions: Other: observation

INTERVENTIONS:
Other: observation — observation

SUMMARY:
The aim of this observational study is to analyze how impaired proprioception affects the gait, reaction time, balance and functioning of stroke patients.

Research questions:

* Are there correlations between the deficit of proprioception and reaction time and the parameters of gait and balance as well as the functional state of stroke patients?
* Are there relationships between factors such as proprioception, reaction time, balance, functional status and gait, and time since stroke, the hemisphere where the stroke occurred, and gender?
* Are there differences in proprioception deficits and reaction times between the lower limbs in stroke survivors?

Participants will be assessed once using standard functional clinical tests and the rehabilitation devices.

Researchers will compare stroke patients and healthy volunteers to see, if there are differences in proprioception deficits, reaction time and balance.

DETAILED DESCRIPTION:
For this prospective observational study, 50 ischemic - stroke survivors (study group) and 50 healthy volunteers matched for age and gender (control group) will be recruited. Study procedures will be performed in the morning including one-time functional assessment of proprioception, gait, balance and reaction time using standard clinical tests (Timed Up and Go Test, sit to stand test, 10m walk test, Wisconsin scale, Berg scale, Ashworth scale, Brunstrom scale, Barthel Scale, Rankin scale and FAC) and rehabilitation devices (Luna EMG - proprioception assessment, Pablo - gait parameters assessment, Omego Plus - proprioception assessment, ALFA stabilometric platform - balance and reaction time assessment).

ELIGIBILITY:
Inclusion Criteria:

* informed and voluntary consent of the patient,
* first-time stroke,
* hemiparesis,
* time from stroke to 3 months,
* age 30-75,
* grade 3-5 in the Functional Ambulation Category,
* walking without orthopedic support.

Exclusion Criteria:

* lack of informed and voluntary consent of the patient,
* second or subsequent stroke,
* stroke of the brainstem and cerebellum,
* epilepsy,
* disorders of higher mental functions,
* coexisting neurological, rheumatological, orthopedic diseases,
* use of orthopedic supplies during locomotion.

Ages: 30 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 50 stroke survivors up to 3 months after the stroke - patients reffered to the Department of Rehabilitation, Clinical Regional Hospital number 2 in Rzeszow, Poland (study group) and 50 healthy volunteers matched for age and gender.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-11-08 (Actual); Primary Completion 2024-09-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Correlation between the knee proprioception deficit (degree) and gait speed (m/s) | September 2024
  The knee proprioception deficit (degree) will be assessed by rehabilitation robot Luna EMG and gait speed (m/s) will be assessed using inertial sensors (Pablo device)
Correlation between the knee proprioception deficit (degree) and gait time: 10-meter-Walk Test (seconds) | September 2024
  The knee proprioception deficit (degree) will be assessed by rehabilitation robot Luna EMG and gait time (seconds) will be assessed using inertial sensors (Pablo device)
Correlation between the knee proprioception deficit (degree) and gait cycle (steps/minute) | September 2024
  The knee proprioception deficit (degree) will be assessed by rehabilitation robot Luna EMG and gait cycle (steps/minute) will be assessed using inertial sensors (Pablo device)
Correlation between the knee proprioception deficit (degree) and cycle distance (cm) | September 2024
  The knee proprioception deficit (degree) will be assessed by rehabilitation robot Luna EMG and cycle distance (cm) will be assessed using inertial sensors (Pablo device)
Correlation between the knee proprioception deficit (degree) and ambulation status: Functional Ambulation Category (points: minimum 0, maximum 5) | September 2024
  The knee proprioception deficit (degree) will be assessed by rehabilitation robot Luna EMG and the ambulation status will be assessed using standard clinical scale: Functional Ambulation Category. Less points indicate worse ambulation category
Correlation between the knee proprioception deficit (degree) and kinematic and spatiotemporal gait parameters: Wisconsin scale (points: minimum 13.35, maximum 42) | September 2024
  The knee proprioception deficit (degree) will be assessed by rehabilitation robot Luna EMG and the kinematic and spatiotemporal gait parameters will be assessed using standard clinical scale: Wisconsin scale. The higher the score the more seriously affected the gait
Correlation between the knee proprioception deficit (degree) and reaction time (miliseconds) | September 2024
  The knee proprioception deficit (degree) will be assessed by rehabilitation robot Luna EMG and the reaction time will be assessed using stabilometric platform (Alfa)
Correlation between the knee proprioception deficit (degree) and balance parameter: lateral sways (cm) | September 2024
  The knee proprioception deficit (degree) will be assessed by rehabilitation robot Luna EMG and the lateral sways (cm) will be assessed using stabilometric platform (Alfa)
Correlation between the knee proprioception deficit (degree) and balance parameter: anterior-posterior sways (cm) | September 2024
  The knee proprioception deficit (degree) will be assessed by rehabilitation robot Luna EMG and the anterior-posterior sways (cm) will be assessed using stabilometric platform (Alfa)
Correlation between the knee proprioception deficit (degree) and balance parameter: path length (cm) | September 2024
  The knee proprioception deficit (degree) will be assessed by rehabilitation robot Luna EMG and the path length (cm) will be assessed using stabilometric platform (Alfa)
Correlation between the knee proprioception deficit (degree) and balance parameter: lateral velocity (cm/s) | September 2024
  The knee proprioception deficit (degree) will be assessed by rehabilitation robot Luna EMG and the lateral velocity (cm/s) will be assessed using stabilometric platform (Alfa)
Correlation between the knee proprioception deficit (degree) and balance parameter: anterio-posterior velocity (cm/s) | September 2024
  The knee proprioception deficit (degree) will be assessed by rehabilitation robot Luna EMG and the anterior-posterior velocity (cm/s) will be assessed using stabilometric platform (Alfa)
Correlation between the knee proprioception deficit (degree) and balance parameter: COP area (cm2) | September 2024
  The knee proprioception deficit (degree) will be assessed by rehabilitation robot Luna EMG and the COP area (cm2) will be assessed using stabilometric platform (Alfa). COP - center of pressure
Correlation between the knee proprioception deficit (degree) and balance: Berg Balance Scale (points: minimum 0, maximum 56) | September 2024
  The knee proprioception deficit (degree) will be assessed by rehabilitation robot Luna EMG and the balance will be assessed using standard clinical scale: Berg Balance Scale. Less points indicate worse balance
Correlation between the knee proprioception deficit (degree) and dynamic balance: Timed Up and Go Test (seconds) | September 2024
  The knee proprioception deficit (degree) will be assessed by rehabilitation robot Luna EMG and the dynamic balance will be assessed using standard clinical scale Timed Up and Go Test. Longer time of performing test indicates worse dynamic balance
Correlation between the knee proprioception deficit (degree) and functional status: 5 times Sit To Stand Test (seconds) | September 2024
  The knee proprioception deficit (degree) will be assessed by rehabilitation robot Luna EMG and the functional status will be assessed using standard clinical scale: 5 times Sit To Stand Test. Longer time of performing test indicates worse functional status
Correlation between the knee proprioception deficit (degree) and spasticity: Modified Ashworth Scale (points: minimum 0, maximum 4) | September 2024
  The knee proprioception deficit (degree) will be assessed by rehabilitation robot Luna EMG and the spasticity will be assessed using standard clinical scale: Modified Ashworth Scale. Better score indicates worse spasticity
Correlation between the knee proprioception deficit (degree) and functional status: Brunnstrom scale (points: minimum 1, maximum 6) | September 2024
  The knee proprioception deficit (degree) will be assessed by rehabilitation robot Luna EMG and the functional status will be assessed using standard clinical scale: Brunnstrom scale. Better score indicates better functional status
Correlation between the knee proprioception deficit (degree) and functional status: Rankin scale (points: minimum 0, maximum 5) | September 2024
  The knee proprioception deficit (degree) will be assessed by rehabilitation robot Luna EMG and the functional status will be assessed using standard clinical scale: Rankin scale. Better score indicates worse functional status
Correlation between the knee proprioception deficit (degree) and functional status: Barthel scale (points: minimum 0, maximum 100) | September 2024
  The knee proprioception deficit (degree) will be assessed by rehabilitation robot Luna EMG and the functional status will be assessed using standard clinical scale: Barthel. Better score indicates better functional status

SECONDARY OUTCOMES:
Differences in knee proprioception deficit (degree). | December 2024
  The knee proprioception deficit (degree) will be assessed by rehabilitation robot Luna EMG
Differences in gait speed (m/s) | December 2024
  Gait speed will be assessed using inertial sensors (Pablo device)
Differences in gait time: 10-meter-Walk Test (seconds) | December 2024
  Gait time will be assessed using inertial sensors (Pablo device)
Differences in gait cycle (steps/minute) | December 2024
  Gait cycle will be assessed using inertial sensors (Pablo device)
Differences in cycle distance (cm) | December 2024
  Cycle distance will be assessed using inertial sensors (Pablo device)
Differences in ambulation status: Functional Ambulation Category (points: minimum 0, maximum 5) | December 2024
  The ambulation status will be assessed using standard clinical scale: Functional Ambulation Category. Less points indicate worse ambulation category
Differences in kinematic and spatiotemporal gait parameters: Wisconsin scale (points: minimum 13.35, maximum 42) | December 2024
  The kinematic and spatiotemporal gait parameters will be assessed using standard clinical scale: Wisconsin scale. The higher the score the more seriously affected the gait
Differences in reaction time (ms). | December 2024
  Reaction time will be assessed using stabilometric platform (Alfa)
Differences in balance parameter: lateral sways (cm) | December 2024
  Lateral sways will be assessed using stabilometric platform (Alfa)
Differences in balance parameter: anterior-posterior sways (cm) | December 2024
  Anterior-posterior sways will be assessed using stabilometric platform (Alfa)
Differences in balance parameter: path length (cm) | December 2024
  Path length will be assessed using stabilometric platform (Alfa)
Differences in balance parameter: lateral velocity (cm/s) | December 2024
  Lateral velocity will be assessed using stabilometric platform (Alfa)
Differences in balance parameter: anterior-posterior velocity (cm/s) | December 2024
  Anterior-posterior velocity will be assessed using stabilometric platform (Alfa)
Differences in balance parameter: COP area (cm2) | December 2024
  This balance parameter will be assessed using stabilometric platform (Alfa); COP - center of pressure
Differences in balance: Berg Balance Scale (points: minimum 0, maximum 56) | December 2024
  Balance will be assessed using standard clinical scale: Berg Balance Scale. Less points indicate worse balance
Differences in dynamic balance: Timed Up and Go Test (seconds) | December 2024
  Dynamic balance will be assessed using standard clinical scale Timed Up and Go Test. Longer time of performing test indicates worse dynamic balance
Differences in functional status: 5 times Sit To Stand Test (seconds) | December 2024
  The functional status will be assessed using standard clinical scale: 5 times Sit To Stand Test. Longer time of performing test indicates worse functional status
Differences in spasticity: Modified Ashworth Scale (points: minimum 0, maximum 4) | December 2024
  The spasticity will be assessed using standard clinical scale: Modified Ashworth Scale. Better score indicates worse spasticity
Differences in functional status: Brunnstrom scale (points: minimum 1, maximum 6) | December 2024
  The functional status will be assessed using standard clinical scale: Brunnstrom scale. Better score indicates better functional status
Differences in functional status: Rankin scale (points: minimum 0, maximum 5) | December 2024
  The functional status will be assessed using standard clinical scale: Rankin scale. Better score indicates worse functional status
Differences in functional status: Barthel scale (points: minimum 0, maximum 100) | December 2024
  The functional status will be assessed using standard clinical scale: Barthel scale. Better score indicates better functional status

CONTACTS AND LOCATIONS:
Overall Officials: Maciej Kochman, Dr., Principal Investigator — Institute of Health Sciences, College of Medical Sciences, University of Rzeszów
Locations (1):
- Department of Rehabilitation, Clinical Regional Hospital number 2, Rzeszów, Podkarpackie Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: Undecided